CLINICAL TRIAL: NCT02571998
Title: A Phase 2, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Multicenter Study to Evaluate the Safety and Efficacy of CLS001 Topical Gel Versus Vehicle Applied Once Daily for 12 Weeks to Female Subjects With Moderate to Severe Acne Vulgaris
Brief Title: A Study to Evaluate the Safety and Efficacy of Omiganan (CLS001) Topical Gel Versus Vehicle in Female Subjects With Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-009
Record Dates: First submitted 2015-10-02; First posted 2015-10-08 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Omiganan; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Omiganan (CLS001) Topical Gel applied once daily
  Interventions: Drug: Omiganan (CLS001) Topical Gel
- Vehicle Gel (Placebo Comparator): Vehicle Topical Gel applied once daily
  Interventions: Drug: Vehicle Topical Gel

INTERVENTIONS:
Drug: Omiganan (CLS001) Topical Gel
  Arms: Treatment
Drug: Vehicle Topical Gel
  Arms: Vehicle Gel

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of Omiganan (CLS001) topical gel compared to vehicle topical gel applied once daily for 12 weeks in female subjects with moderate to severe inflammatory acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant female subjects ≥ 12 years of age with facial acne vulgaris
* Subjects with an Investigator's Global Assessment (IGA) of Inflammatory Lesions of Acne Vulgaris of Moderate (3) or Severe (4) at Baseline.
* Subjects with ≥ 30 facial inflammatory lesions

Exclusion Criteria:

* Subjects with < 10 or > 75 facial non-inflammatory lesions
* Subjects with > 3 facial nodular or cystic lesions at Baseline
* Standard exclusion criteria

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in inflammatory lesion counts at week 12 | 12 weeks

SECONDARY OUTCOMES:
Absolute change from Baseline at each visit in inflammatory lesions, non-inflammatory lesions, and total lesions | 12 weeks
Percentage of subjects with at least a two grade reduction in the IGA of Inflammatory Lesions of Acne Vulgaris at each visit | 12 weeks
Percentage of subjects with an IGA of Inflammatory Lesions of Acne Vulgaris of clear or almost clear (0 or 1) at each visit | 12 weeks
Percentage of subjects with an IGA of Inflammatory Lesions of Acne Vulgaris of clear or almost clear (0 or 1) and at least a two grade reduction in the IGA of Inflammatory Lesions of Acne Vulgaris at each visit. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Santa Ana, California
  - Santa Monica, California
  - Denver, Colorado
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Miami, Florida
  - Pinellas Park, Florida
  - Sanford, Florida
  - Tampa, Florida
  - Beverly, Massachusetts
  - Fort Gratiot, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Newington, New Hampshire
  - Albuquerque, New Mexico
  - New York, New York
  - Stony Brook, New York
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Knoxville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Pflugerville, Texas
  - San Antonio, Texas
  - Webster, Texas
  - Salt Lake City, Utah
  - Spokane, Washington